CLINICAL TRIAL: NCT01455324
Title: Evaluation of the Development of an Advanced, Conformable Prosthetic Socket, Study II
Status: Completed | Type: Observational
Sponsor: Infoscitex Corporation (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kristen Leroy, Group Leader, Biomedical Devices, Infoscitex Corporation
Other Study IDs: IST1288 Study 2; W81XWH-07-C-0094 (Other Grant/Funding Number: US Army MRMC)
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Evaluation of a New Prosthetic Socket Liner Material
Keywords: prosthetic socket; residual limb volume fluctuation; conformable socket liner

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lower Limb Amputees: Those with lower limb amputations
  Interventions: Device: Novel conformable woven inner socket

INTERVENTIONS:
Device: Novel conformable woven inner socket — Prosthetic socket liner fabricated from novel materials to allow passive conformability for the user

SUMMARY:
The purpose of this study is to work with prosthetists to fit the novel conformable socket material developed by Infoscitex, to subjects, and determine if it is a viable alternative to current prosthetic socket liners. During this task, the research team will travel to the prosthetists locations to have them fit the subject with the conformable woven socket and a check socket, and provide subjective feedback with regard to comfort and fit for the amputee, its ease of use, and breathability. The subject will also wear the woven socket for gait analysis and provide his/her feedback as well.

DETAILED DESCRIPTION:
Modern prosthetics have improved significantly with regards to control and functionality, but the fit of the residual limb within a prosthetic socket is a primary concern for many amputees. A poor fit can lead to skin irritation, tissue breakdown, and pain. The volume of the residual limb of an amputee changes throughout the course of a day and throughout the year. Volume fluctuation within the socket can lead to issues for the amputee, including decreased comfort, increased shear forces, increased pressure on bony prominences, as well as a poor gait pattern. An uncomfortable or non-performing socket/residual limb interface decreases user compliance with the prosthetic and therefore decreases the activity level of amputees who want to remain active in their civilian and military lives. The investigators are developing a multilayered socket that takes advantage of a novel braided material for strength and passive conformability with thin layers dedicated to wearer comfort. This new socket provides ultimate fit for improvement in the performance of the prosthesis. The socket adapts itself to the changing physical shape of the residual limb as the prosthesis is worn. The adaptation is a natural result of the material properties, so is done passively and in real time. The materials are lightweight, breathable, and ultrasound transparent, allowing the prosthetic to function in a variety of environments.

This study will be undertaken to have prosthetists fit subject lower limb amputees with the woven inner socket, with a check socket for evaluation in a gait lab setting. At the completion, the subject and prosthetists will be asked to complete a questionnaire and give their opinions regarding the material of the woven inner socket.

ELIGIBILITY:
Inclusion Criteria:

* lower limb amputation
* stable residual limb volume
* loss of limb due to trauma
* at least 18 years of age

Exclusion Criteria:

* evidence or history of neuropathy
* presence of phantom limb pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject will be selected from one prosthetic fabrication facility and recruited by their prosthetist
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States